CLINICAL TRIAL: NCT01828086
Title: A Randomized, Double-blind, Placebo and Positive Controlled, Single and Multiple Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CJM112 in Chronic Plaque-type Psoriasis Patients
Brief Title: Single and Multiple Dose Escalation Study to Assess the Safety and Tolerability of CJM112 in Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCJM112X2101
Record Dates: First submitted 2013-04-05; First posted 2013-04-10 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2019-03

CONDITIONS: Chronic Plaque-type Psoriasis
Keywords: Psoriasis, chronic plaque-type psoriasis, IL17, monoclonal antibody
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CJM112 (Experimental): CJM112 in different doses; single ascending and multiple ascending
  Interventions: Biological: CJM112
- Placebo (Placebo Comparator): Placebo to match
  Interventions: Other: Placebo
- Secukinumab (Active Comparator): Active investigational drug.
  Interventions: Biological: Secukinumab

INTERVENTIONS:
Biological: CJM112 — Monoclonal antibody
  Arms: CJM112
Biological: Secukinumab — Monoclonal antibody
  Other Names: AIN475
  Arms: Secukinumab
Other: Placebo — Liquid for subcutaneous injection without active drug.
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo and positive controlled, single and multiple dose study to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of CJM112 in chronic plaque-type psoriasis patients. This trial never made it to the Phase II part of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18-65 years of age at time of consent
* Chronic plaque-type psoriasis diagnosed for at least 6 months at time of randomization
* At randomization, moderate to severe psoriasis as defined by:
* PASI score of 12 or greater and,
* IGA score of 3 or greater and,
* Body Surface Area (BSA) affected by plaque-type psoriasis of 10% or greater.
* Female patients may be included according to the following:

Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, using highly effective methods of contraception during dosing and for 5 times the terminal half-life of study treatment.

• Male subjects must agree to comply with two highly effective contraceptive methods

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type (incl. drug induced psoriasis)
* Ongoing use of prohibited psoriasis treatments and other prohibited medication at randomization. Washout periods detailed in the protocol have to be adhered to
* Previous treatment with IL-17 or IL17R blocking agents, including secukinumab
* Any live vaccines (including nasal-spray flu vaccine) starting from 6 weeks before screening, during the study, and up to 24 weeks after the last dose of CJM112 or secukinumab
* Evidence of active tuberculosis at screening
* Active systemic infections (other than common cold)
* Pregnant or nursing (lactating) women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety | 19 weeks
  Safety as assessed by the number of participants with adverse events as measured by laboratory parameters, vital signs, electrocardiogram and the collection of serious and non-serious adverse events.

SECONDARY OUTCOMES:
Psoriasis Area and Severity Index (PASI) | 19 weeks
Total CJM112 Concentrations in Serum | 19 weeks
  Measurement of drug levels in the blood of treated patients.
Concentration of anti-CJM112 Antibodies in Serum | 19 weeks
  Assessment of the ability of the compound to evoke an immune response. Assessed in blood of treated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- United States (17):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Encino, California
  - Novartis Investigative Site, North Hollywood, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Normal, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Crowley, Louisiana
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CCJM112X2101 from the Novartis Trial Results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=15349
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=36